CLINICAL TRIAL: NCT02131831
Title: Telomeres Parameters in Cirrhosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, ido laish, phsician in gastroenterology institute, Meir Medical Center
Other Study IDs: IDO 123 TRX
Record Dates: First submitted 2014-04-26; First posted 2014-05-06 (Estimated); Last update posted 2014-09-16 (Estimated); Status verified 2014-09

CONDITIONS: Cirrhosis
Keywords: telomere; telomerase; cirrhosis
MeSH Terms: conditions — Fibrosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood

GROUPS / COHORTS (1):
- cirrhosis

SUMMARY:
There are several factors that influence telomere length in patients with cirrhosis, such as metabolic derangements and infectious etiologies, The aim of the study is to compare telomere length and other parameters related to genetic instability in telomere/ telomerase system, in peripheral blood lymphocytes in cirrhosis from different etiologies.

ELIGIBILITY:
Inclusion Criteria:

* cirrhotic patients from different etiologies

Exclusion Criteria:

* decompensated cirrhosis (Child C)
* age under 18 years
* any known malignancy, including hepatocellular carcinoma
* patient that are unable to sign for informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with cirrhosis
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2014-06; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
telomerase activity | baseline
  number of copies of telomerase in peripheral blood lymphocytes, as determined by FISH

CONTACTS AND LOCATIONS:
Locations (1):
- Meir Medical Center, Kfar Saba, Israel